CLINICAL TRIAL: NCT03095768
Title: Blending Lifestyle Education and Nutrition Demonstration for Seniors in the Warrensville Heights Community
Brief Title: Lifestyle Education and Nutrition Demonstration
Acronym: BLENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: City of Warrensville Heights (Unknown); Ohio Department of Aging (Unknown)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-046
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Chronic Disease
Keywords: Lifestyle; Nutrition; Cooking
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Lifestyle Education and Cooking Demonstration
  Interventions: Other: Lifestyle Education and Cooking Demonstration

INTERVENTIONS:
Other: Lifestyle Education and Cooking Demonstration — Participants will receive an interactive cooking demonstration as well as healthy lifestyle education

SUMMARY:
The Center for Lifestyle Medicine at the Cleveland Clinic Wellness Institute has a proven track record of engaging patients in healthy living and eating through education, live cooking demonstrations / hands-on cooking classes, exercise and stress management programs.

As a result of the Community Health Needs Assessment, we are collaborating with Cleveland Clinic Community Outreach and 12th District Representative, John E. Barnes, Jr., to extend our expertise to the community of Warrensville Heights, Ohio.

DETAILED DESCRIPTION:
The City of Warrensville Heights and The Cleveland Clinic are combining efforts to address the paucity of fresh and nutritious foods accessible to seniors in the Warrensville Heights community through a new program at the city's Civic and Senior Center. This program will combine healthy lifestyle education with nutrition demonstration using recipes that can be prepared in a blender. These recipes have been designed to be simple, delicious and easy to eat, and include smoothies, soups and even a few desserts! Our ultimate goal is to use both education and demonstration to promote a mindset change regarding community members' abilities to eat healthy.

The population in the Warrensville Heights community is aging, and there is a high prevalence of chronic diseases including hypertension, diabetes, obesity and kidney disease. A recent Community Health Needs Assessment (CHNA) identified engagement and participation in the promotion and maintenance of a healthy lifestyle as a major area for improvement. Currently there is very limited access to healthy foods in the immediate community of Warrensville Heights, and in many cases, the transportation costs required for residents to access those healthy foods is often financially unfeasible. It is clear from this CHNA that both access to and education about healthy food options is sorely needed in this community.

The Center for Lifestyle Medicine at the Cleveland Clinic Wellness Institute has a proven track record of engaging patients in healthy living and eating through education, live cooking demonstrations / hands-on cooking classes, exercise and stress management programs. In response to the CHNA and in collaboration with 12th District Representative, John E. Barnes, Jr., the BLENDS study will extend our expertise to the Warrensville Heights community.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 55 years of age or older living in the neighborhoods of Warrensville Heights

Exclusion Criteria:

1. Food allergies
2. Celiac or non-Celiac gluten intolerance
3. Travel plans that do not permit full participation in the intervention
4. Recent unexplained weight loss (10 pounds or more in past 3 months)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Behavior Change from Baseline to 2 Months | 2 months
  Food Frequency Surveys

SECONDARY OUTCOMES:
Change from Baseline BMI at 2 Months | 2 months
  Body Mass Index (kg/m^2)
Change from Baseline Waist Circumference at 2 Months | 2 months
  Waist Circumference (cm)
Change from Baseline Blood Pressure at 2 Months | 2 months
  Blood Pressure (mmHg)
Change from Baseline Glucose at 2 Months | 2 months
  Point-of-care Glucose (mg/dL)
Change from Baseline Cholesterol at 2 Months | 2 months
  Point-of-care Cholesterol (mmol/L)
Change in Quality of Life from Baseline to 2 Months | 2 months
  SF-36 Survey
Program Evaluation Survey | 2 months
  Investigator-created Survey

CONTACTS AND LOCATIONS:
Overall Officials: Dana L Schneeberger, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Warrensville Heights Senior Center, Warrensville Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No